CLINICAL TRIAL: NCT06829056
Title: Presence of Pain Shows Greater Effect Than Tendon Structural Alignment During Landing Dynamics
Status: Completed | Type: Observational
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Collaborators: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Daniela Ferreira Carneiro, Master's degree in Physiotherapy, Escola Superior de Tecnologia da Saúde do Porto
Other Study IDs: FIS-2022-06
Record Dates: First submitted 2025-02-10; First posted 2025-02-17 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Patellar Tendon; Athletes
Keywords: jump performance; patellar tendon; tendon structure; UTC

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Athletes: Included volunteer participants were aged between 18-30 years, competing in the highest-level Portuguese volleyball league with a minimum of 10 years of volleyball practice. Participants were excluded in presence of injuries or discomfort that impeded maxi- mal jumping tests, history of surgery within the last 12 months or illness during data collection.

SUMMARY:
The goal of this observational study is to investigate the relationship between temporal, kinetic, and kinematic jump variables and patellar tendons' structure in athletes. The main research questions are:

Does the structure of the patellar tendon relate to the temporal, kinetic, and kinematic variables of different jumps?

To answer these questions, participants will undergo a UTC (Ultrasound Tissue Characterization) scan of the patellar tendon and perform two vertical jump: a countermovement jump and tuck jump test.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18-30 years;
* competing in the highest-level Portuguese volleyball league with a minimum of 10 years of volleyball practice.

Exclusion Criteria:

* presence of injuries or discomfort that impeded maximal jumping tests;
* history of surgery within the last 12 months;
* illness during data collection

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The target population for this study consisted of volleyball athletes aged 18 to 35, of both sexes.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Tendon Structure | Baseline
  Ultrasound Tissue Characterization (UTC) captures tendon structure and quantifies the number of altered fibers. This technology classifies tendon structure into four echo types, reflecting tendon integrity and fibrillar organization. Data collection for the patellar tendon will be conducted with participants seated, hips and knees at 90° flexion, and feet supported on a stable surface. For the Achilles tendon, the participants will be lying down with ankle in neutral position. This positioning ensures the probe is aligned transversely to the tendons, enabling the acquisition of optimal ultrasound images without anisotropy. Ultrasound parameters will be standardized for all scans: a 40-second B-mode ultrasound using a 7-10 Hz linear transducer, with the probe attached to a tracking device that moves automatically along the tendon's perpendicular axis, capturing consecutive images at 0.2 mm intervals. A single scan of the tendons will be performed for each knee.
Jump Variables | baseline
  The data collection protocol includes the following tasks: countermovement jump and tuck jump test. Kinematic variables will be analyzed by recording the spatial positions of reflective markers placed on specific anatomical regions. Data will be captured using the Qualisys Motion Capture System (version 2021.2). Ground reaction forces will be measured using a force platform connected to a signal amplifier. The platform records the three components of ground reaction forces-anteroposterior, mediolateral, and vertical-via four sensors. The image capture hardware is connected to the Qualisys USB Analog Acquisition interface, synchronizing temporal, kinetic, and kinematic data with the Qualisys Track Manager (QTM) software.

CONTACTS AND LOCATIONS:
Locations (1):
- Escola Superior de Saúde do Instituto Politécnico do Porto, Porto, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No